CLINICAL TRIAL: NCT06543225
Title: Awareness Of Gynecologists About Role Of Physical Therapy In Management Of Polycystic Ovarian Syndrome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rolan Khaled Kamal El Dein, Principal investigator, Cairo University
Other Study IDs: PT REC/012/004408
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: poly cystic ovarian syndrome
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Egyptian Gynecologists: Egyptian gynecologists were included in the study to determine their awareness about the role of physiotherapists in the treatment of PCOS.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aimed to measure the extent of knowledge of gynecologists about the role of physical therapy in the management of PCOS.

DETAILED DESCRIPTION:
Physical therapists are good communicators and also have the knowledge and skills to make a substantial impact in this field of management of polycystic ovarian syndrome.

It is important for the gynecologists to have awareness about the role of physical therapy in polycystic ovarian syndrome to encourage patient to seek physical therapy help instead of suffering in silence and improve their quality of life

ELIGIBILITY:
Inclusion Criteria:

* Gynecologists with more than 2 years' experience.
* Had managed cases of PCOS.

Exclusion Criteria:

* Gynecologists with less than 2 years' experience.
* Gynecologists who didn't deal with PCOS.

Ages: 29 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian gynecologists were included in the study to determine their awareness about the role of physiotherapists in the treatment of PCOS.
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Awareness and knowledge of gynecologists about role of physiotherapists in the treatment of PCOS | 8 months
  A specially designed questionnaire was used to identify the awareness and knowledge of gynecologists about the physiotherapy role in the treatment of PCOS

CONTACTS AND LOCATIONS:
Overall Officials: Soheir EL-Kosery, professor, Study Chair — Cairo University
Locations (1):
- Rolan Khaled Kamal El Dein, Tanta, El Gharbia, Egypt